CLINICAL TRIAL: NCT01830361
Title: A Single-arm Phase II Trial to Assess the Efficacy of Midostaurin (PKC412) Added to Standard Primary Therapy in Patients With Newly Diagnosed c-KIT or FLT3-ITD Mutated t(8;21) AML
Brief Title: Trial to Assess the Efficacy of Midostaurin (PKC412) in Patients With c-KIT or FLT3-ITD Mutated t(8;21) AML
Acronym: MIDOKIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-MIDOKI-052; 2011-002567-17 (EudraCT Number)
Record Dates: First submitted 2013-03-25; First posted 2013-04-12 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; c-KIT; FLT3-ITD; t(8;21); chemotherapy; midostaurin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- midostaurin (PKC412), capsules (Experimental): midostaurin 50 mg (two 25 mg capsules) is given in combination with the second of two induction cycles and in combination with three cycles of high-dose cytarabine (HiDAC) consolidation chemotherapies and maintenance treatment in patients with c-kit or FLT3-ITD positive t(8;21) AML in an open-label one-arm design. The first cycle of induction is not part of the study.
  Interventions: Drug: midostaurin (PKC412)

INTERVENTIONS:
Drug: midostaurin (PKC412) — Midostaurin 50 mg (2 capsules) twice daily days 8-21 in induction II + consolidation I-III; maintenance treatment twice daily continuously for 12 months
  Other Names: Rydapt

SUMMARY:
To assess the efficacy of tyrosine-kinase inhibitor midostaurin in c-KIT or FLT3-ITD mutated t(8;21) AML. To assess the efficacy of midostaurin depending on the type of c-KIT mutation

DETAILED DESCRIPTION:
AML patients displaying t(8;21) have a relatively favourable outcome. Nevertheless, only approximately 50% of patients carrying this cytogenetic aberration are alive at 5 years. This suggests that some patients have more aggressive leukemic phenotypes and indicates the need for treatment optimization with novel therapies.

The mutated KIT gene as well as the FLT3-ITD mutation have recently been identified as factors most likely to explain the heterogeneous clinical outcomes within the group of t(8;21) AML. The FLT3 and c-KIT genes encode type III receptor tyrosine kinases (RTK) with important and partly redundant functions in early hematopoietic stem cells. Various activating mutations have been described for both genes. For c-KIT, the incidence ranges from 17 to 48% depending on the source population and type of mutations determined. It has been consistently shown that in AMLs with t(8;21), mutated c-KIT is associated with a dramatically increased risk of relapse and reduced overall survival compared to their unmutated counterparts. The FLT3-ITD mutation has a similar negative effect on prognosis in the patient group of t(8;21) mutated AMLs as c-KIT.

PKC412 (midostaurin) is known to inhibit the c-KIT RTK activity as well as the FLT3 kinase, both in patients with ITD and TKD mutations. It should therefore be possible to abrogate the negative impact of pathologically increased c-KIT or FLT3-ITD activity on relapse and overall survival by using midostaurin in this patient population. Aim of the proposed clinical trial is to prove the efficacy of midostaurin in c-KIT or FLT3-ITD mutated t(8;21)- AMLs in an open-label one-arm design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of c-KIT mutated t(8;21) AML i.e.

  1. >20% myeloid blasts in bone marrow and/or peripheral blood at initial diagnosis
  2. Plus cytogenetic diagnosis of aberration t(8;21)/AML1-ETO
  3. Plus mutation of c-KIT gene (mut-KIT17 or mut-KIT8) or FLT3-ITD mutation or both c-KIT and FLT3-ITD mutations
* Chemoresponsive disease as determined by early bone marrow assessment on day 14-16 after first cycle of induction therapy with cytarabine in combination with daunorubicine or idarubicine, or mitoxantrone- Fit for further intensive chemotherapy
* Age 18-65 years
* ECOG performance status of 0-2
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Primary refractory or previously relapsed AML
* Non-eligibility for high-dose cytarabine based consolidation, e.g. intolerance to cytarabine
* Inability to swallow oral medications
* Symptomatic congestive heart failure
* Bilirubin >2.5 x upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Event-free Survival | 2-year Event-free Survival

SECONDARY OUTCOMES:
Time to relapse | 2-years
Overall survival | 2-years
Relapse-free survival | 2-years
morphologic and molecular CR rate | 2-years
incidence of AEs/SAEs | until 30 days after end of treatment
MRD kinetics (molecular residual disease) | 2-years
  molecular diagnostics of markers in peripheral blood / bone marrow
Cumulative incidence of relapse | 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof. Dr., Principal Investigator — Medizinische Fakultät der TU Dresden, Medizinische Klinik und Poliklinik I
Locations (10):
- Germany (10):
  - Klinikum Chemnitz gGmbH, Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum Dresden Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Erlangen, Medizinische Klinik 5, Erlangen
  - Klinikum der Johann-Wolfgang-Goethe Universität, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Universitätsklinikum Münster, Münster
  - Städtisches Klinikum Nord, Nuremberg
  - Klinikum der Universität Regensburg, Regensburg

REFERENCES:
- See also: Website Study Alliance Leukemia (coordinating study group) — http://www.sal-aml.org